CLINICAL TRIAL: NCT06448949
Title: Hemodynamic Study of In-Stent Stenosis After Flow Diverter Implantation for Intracranial Aneurysms Based on 3D-DSA Combined With TCCD
Brief Title: Hemodynamic Study of In-Stent Stenosis(I) After Flow Diverter(F) Based on 3D-DSA(D) Combined With TCCD(T)
Acronym: DTFI
Status: Recruiting | Type: Observational
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: LC20240520
Record Dates: First submitted 2024-06-03; First posted 2024-06-07 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Hemodynamics;In-stent Stenosis;Transcranial Doppler;Intracranial Aneurysm;Flow Diverter; Prospective Cohort Study
Keywords: Hemodynamics.in-stent stenosis.Transcranial Doppler.Intracranial Aneurysm.flow diverter.Prospective cohort study.Mechanical thrombectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TB and PED
  Interventions: Other: Flow Diverter Implantation

INTERVENTIONS:
Other: Flow Diverter Implantation — Patients must undergo flow diverter implantation and have DSA examinations of the parent artery and TCCD examinations of Flow Diverter Implantation performed preoperatively, three days postoperatively, and six months postoperatively.

SUMMARY:
DTFI is a single-center, prospective cohort study aimed at evaluating the hemodynamics of in-stent stenosis after flow diverter implantation, seeking to identify the threshold effect of blood flow in stenosis.

DETAILED DESCRIPTION:
DTFI study investigates the hemodynamic changes in patients with intracranial aneurysms who have undergone flow diverter implantation, using a combination of three-dimensional digital subtraction angiography (3D-DSA) and transcranial color-coded duplex (TCCD) sonography. The aim is to understand the development of in-stent stenosis and its impact on blood flow.

ELIGIBILITY:
Inclusion Criteria:

Age ≥ 18, male or non-pregnant female. Diagnosis of intracranial aneurysm confirmed by DSA (Digital Subtraction Angiography).

Intracranial aneurysms treated with flow diverter (FD). DSA follow-up of at least 1 month.

Exclusion Criteria:

Secondary intracranial aneurysm cases: traumatic aneurysms, infectious aneurysms, or aneurysms associated with arteriovenous malformations (AVM) or vasculitis.

Previously treated recurrent aneurysm or target aneurysm with craniotomy clipping surgery or other endovascular interventions.

Aneurysms located at the distal end of the circle of Willis where TCCD (Transcranial Color-Coded Doppler) cannot be detected.

Known familial clustering history. Expected survival less than 1 year. Preoperative clinical assessment with mRS (Modified Rankin Scale) score ≥ 3. Known allergy or contraindication to antiplatelet drugs, anticoagulants, contrast agents, anesthetics, nitinol memory alloy, platinum-tungsten alloy, or platinum-iridium alloy.

Severe respiratory, hepatic, or renal disease (e.g., creatinine ≥ 3.0 mg/dL excluding dialysis) or coagulation disorders.

Undergoing major surgery (e.g., limb fracture fixation, tumor resection, major organ surgery, etc.) within 30 days prior to signing informed consent or planned within 60 days after signing informed consent.

Pregnant or lactating women, or women with a positive pregnancy test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated in the Department of Neurovascular Surgery, Zhujiang Hospital, Southern Medical University, who were confirmed by DSA to have intracranial aneurysms and underwent treatment with FD (flow diverter) implantation.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
operative Hemodynamic Differences ### Pre- and Post-operative Hemodynamic Differences ### Pre- and Post-operative Hemodynamic Differences ### Pre- and Post-operative Hemodynamic Differences ### Pre- and Post-operative Hemodynamic | Preoperatively, 3 days postoperatively, and 6 months postoperatively
  Transcranial Color-Coded Doppler (TCCD) measurements of blood flow velocity
Hemodynamic changes in-stent stenosis | Preoperatively, 3 days postoperatively, and 6 months postoperatively
  Transcranial Color-Coded Doppler (TCCD) measurements of blood flow velocity
The occlusion rate of the aneurysm | 6 months
  The occlusion rate of the aneurysm at 6 months
Proportion of patients without disability at 6 months | 6 months
  mRS score 0-1
Proportion of patients with functional independence at 6 months | 6 months
  mRS score 0-2
Proportion of patients with Symptomatic intracranial hemorrhage(sICH) within 48 hours | Within 48 hours
  ICH will be evaluated according to the Heidelberg Bleeding Classification. sICH is diagnosed if the new observed ICH is associated with any of the following conditions: 1) NIHSS score increased more than 4 points than that immediately before worsening; 2) NIHSS score increased more than 2 points in one category; 3) Deterioration led to intubation, hemicraniectomy, external ventricular drain placement or any other major interventions. Additionally, the symptom deteriorations could not be explained by causes other than the observed ICH.
Incidence of serious adverse events | Within 1 years
  Including but not limited to acute respiratory failure, severe or malignant cerebral artery infarction, acute heart failure, debridement decompression, and other major medical events that can result in death, immediately life-threatening, hospitalization or prolongation of this hospitalization, terminally or severely disabling/incapacitating, the loss of a significant ability to maintain normal life functioning, or medical intervention to avoid the above outcomes.
Procedure-related complications Procedure-related complications | Up to 24 hours
  such as arterial perforation, iatrogenic arterial dissection, embolization in previously uninvolved vascular territory, arterial access site hematoma, and retroperitoneal hematoma. Arterial perforation will be defined at angiography by the operator and associated with subarachnoid hemorrhage. Iatrogenic arterial dissection will be defined at angiography by the operator. Arterial access site hematoma will be assessed as a complication of arterial access puncture and defined by clinical examination and anatomic imaging. Retroperitoneal hematoma will be assessed as a complication of groin puncture and defined by imaging (ultrasound or CT or MR angiography). The definition of embolization in previously uninvolved vascular territory is noted after recanalization of the primary occlusion site, any vessel occlusions distal from the primary occlusion site are considered emboli due to periprocedural thrombus fragmentation.

CONTACTS AND LOCATIONS:
Overall Officials: Duan Chuan zhi, MD, Principal Investigator — Study Principal Investigator
Locations (1):
- DuanChuanzhi, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No